CLINICAL TRIAL: NCT05898932
Title: Enhanced Clinical Decisions for Management of Benign Prostatic Hyperplasia Using Patient-Reported Outcomes
Status: Recruiting | Type: Observational
Sponsor: Northwestern University (Other)
Collaborators: Endeavor Health (Other); University of Chicago (Other)
Responsible Party: Principal Investigator, James W Griffith, Professor, University of Chicago
Other Study IDs: STU00217126
Record Dates: First submitted 2023-05-16; First posted 2023-06-12 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: PROs; Questionnaires; Benign Prostatic Hyperplasia; Lower Urinary Tract Symptoms; BPH; LUTS; Patient reported outcome measures
MeSH Terms: conditions — Prostatic Hyperplasia; Lower Urinary Tract Symptoms | interventions — Practice Management, Medical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Participants will have the option to consent to contributing to a biobank, which would contain DNA and other specimens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Medical Management: Participants will be managing condition with medication
  Interventions: Other: Medical Management
- Surgical Management: Participants will be managing condition with a surgery
  Interventions: Other: Surgical Management

INTERVENTIONS:
Other: Medical Management — Participants will be managing condition with medication
  Groups: Medical Management
Other: Surgical Management — Participants will be managing condition with a surgery
  Groups: Surgical Management

SUMMARY:
The goal of this project is to use newly developed patient-reported outcomes to improve the clinical care of patients with benign prostatic hyperplasia. The use of new patient-centered tools will improve evaluation and clinical decision-making by including symptoms not commonly measured in men, such as urinary incontinence, and allow for more frequent assessment of lower urinary tract symptoms through remote surveillance. Through the use of care-coordination checklists, clinicians can be more responsive to post-treatment symptom changes, resulting in reduced bother from lower urinary tract symptoms and higher quality of life in patients with benign prostatic hyperplasia.

DETAILED DESCRIPTION:
The American Urological Association Symptom Index (AUA-SI) has been the primary patient-reported outcome (PRO) used in men with benign prostatic hyperplasia (BPH) for decades. New symptom indices - the LURN SI-10 and LURN SI-29 - have been developed by the Symptoms of Lower Urinary Tract Dysfunction Research Network (LURN) to provide a general-use multidimensional symptom assessment in the urology clinic. These tools are relatively new and have yet to be validated in specific disease populations. The overarching goal of this project is to use these new questionnaires to enhance clinical decision-making in men with BPH. This will be achieved by (1) integration of PRO assessments into the evaluation and management of patients with BPH; (2) determination of clinical meaningful differences in LURN symptom indices in men with BPH receiving known effective treatment; and (3) creation of data visualization tools and care-coordination recommendations to facilitate the matching of evidence-based treatments to patients with persistent symptoms using PROs. PROs provide a cost-effective remote management strategy that, combined with advances in electronic medical health record technology, can improve patient care by allowing for more real-time surveillance and intervention, and the monitoring of common comorbid symptoms such as sleep disturbance and depression, in addition to core urologic symptoms of BPH.

In Aim 1, the investigators will use sophisticated statistical methods to predict changes in urological symptoms and assess associations between lower urinary tract symptoms and measures of sleep, depression, and pain, among others. In Aim 2, the investigators will assess test-retest reliability and other psychometric properties of the LURN symptom indices, using a triangulation of methods to determine minimally important differences. Finally in Aim 3, the investigators will engage stakeholders, including patients and clinicians, and use qualitative methods to create visualization tools and care coordination checklists to improve counseling and follow up for patients undergoing treatment. Aim 3 will also enhance the recovery and routine monitoring of men with BPH after surgery, who can experience distressing side effects and complications such as urinary leakage and pain.

ELIGIBILITY:
Inclusion Criteria:

1. Male sex
2. Age 50 years or older
3. Diagnosed by physician with BPH
4. Able and willing to complete questionnaires
5. Able and willing to provide informed consent
6. Ability to read, write, and speak in English
7. No plans to move from study area in next 6 months

Exclusion Criteria:

1. Female sex or intersex
2. Younger than 50 years of age
3. Being a prisoner or detainee
4. Gross hematuria
5. Interstitial cystitis
6. Pelvic or endoscopic genitourinary surgery within the preceding 6 months (not including diagnostic cystoscopy)
7. History of cystitis caused by tuberculosis, radiation therapy, or Cytoxan/cyclophosphamide therapy
8. Ongoing symptomatic urethral stricture
9. Current chemotherapy or other cancer therapy
10. History of lower urinary tract or pelvic malignancy
11. Severe neurological of psychiatric disorder that would prevent study participation (e.g., bipolar disorder, psychotic disorder, Alzheimer's Disease)
12. Current moderate or severe substance use disorder

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men with benign prostatic hyperplasia
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Patient rating of global change | Through study completion, from week 4 to week 24
  This is a single item that captures how much better or worse the person's bladder condition is relative to when they began treatment for BPH. The Patient Global Rating of Change (PGRC) scale ranges from "Very much worse" (1) to "Very much improved" (7), with higher scores indicating a better outcome.
LURN SYMPTOM INDEX-29 (LURN SI-29) | The past 7 days
  This is a multidimensional questionnaire that assesses different lower urinary tract symptoms as well as single item about global bother.
The Patient-Reported Outcomes Measurement Information System (PROMIS-29) Profile v2.1 | The past 7 days
  The PROMIS-29 Profile-a 29-item instrument-combines short assessments of eight core constructs of health-related quality of life (HRQoL): physical function (PF), sleep disturbance (SD), pain interference (PI) and pain intensity (PIN), fatigue (FA), anxiety (AN), depression (DE) and ability to participate in social roles and activities (SRAA). PROMIS employs a T-score, which is constructed such that 50 is the mean of the general population, and the standard deviation is 10 by definition. Most scores falling between 20 and 80, which is +/- 3 SDs around the mean. Higher scores represent more of a domain. Therefore, for physical function, higher scores represent better health whereas for anxiety, higher scores represent poorer health.
AMERICAN UROLOGICAL ASSOCIATION (AUS) SYMPTOM SCORE | The past 30 days
  This is a 7-item self-report measure used to assess urinary urgency, frequency, and voiding symptoms. ranges from 0 to 35, with higher scores indicating more severe urinary symptoms.

SECONDARY OUTCOMES:
Sexual Health Inventory for Men (SHIM) Questionnaire | The past 6 months
  This is an instrument widely used measure of erectile function consisting of 5 questions. The severity of erectile dysfunction score is from 1 to 25, with 1 being the most severe and 25 being healthy.
The Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.0 - Gastrointestinal Diarrhea 6a | In the past 7 days
  This contains items focused on capturing the frequency, form, bothersomeness, impact, controllability, and predictability of bowel urgency during the past 7 days. PROMIS employs a T-score, which ranges from 0 to 100, with most scores falling between 20 and 80.Higher scores represent more of a domain
The Patient-Reported Outcomes Measurement Information System (PROMIS) Scale v1.0 - Gastrointestinal Constipation 9a | In the past 7 days
  This assesses the frequency and intensity of incomplete evacuation, rectal pain, straining, and hard stools, as well as the need for manual extraction of stool. PROMIS employs a T-score, which ranges from 0 to 100, with most scores falling between 20 and 80. Higher scores represent more of a domain.
Male Sexual Health Questionnaire for Ejaculatory Dysfunction (MSHQ-EjD) | In the past month.
  A 4-item validated questionnaire used to assess ejaculatory dysfunction. Three questions relate to ejaculatory function items and 1 relates to ejaculation bother item. Ejaculatory function score is the sum of questions 1 to 3 and scores range from 1 to 15, with lower scores indicating more severe ejaculatory complaints. Bother score range from 0 to 5, with higher scores indicating greater bother
The snoring, tiredness, observed apnea, high BP, BMI, age, neck circumference, and male gender (STOP-Bang) questionnaire | Not Applicable (NA)
  The STOP-Bang questionnaire is a scoring model consisting of eight easily administered questions starting with the acronym STOP-Bang (Appendix) and is scored based on Yes/No answers (score: 1/0). Thus, the scores range from a value of 0 to 8. Higher score indicating worse outcome.
3-Day Voiding Diary | Recorded on three separate days
  The diary records the patient's daily fluid intake, frequency of urination throughout the day and night, instances of leakage, and the quantity of lost urine. Analyzing these findings against the standard criteria for regular bladder function could reveal potential issues and help confirm a diagnosis. The definition of normal benchmarks takes into account factors like age, gender, as well as various internal and external variables including fluid consumption and its nature.
The National Cancer Institute (NCI) Quick Food Scan | in the past 12 months
  National Cancer Institute Quick Food Scan estimates fat intake as a percentage of total energy. Participants rate their frequency of consuming 15 food groups and reduced-fat butter or margarine over the last 12 months ranging 1 = never to 8 = more than once per day. Reduced-fat margarine usage as a replacement for butter is rated separately. Scoring is based on weighted least-squares estimates of regression coefficients for data from the U.S. Department of Agriculture's 1994-1996 Continuing Survey of Food Intakes by Individuals. The algorithm accounts for food frequency with age- and sex-specific portion sizes. The final score is expressed as total estimated percentage of dietary energy from fat.
The Patient-Reported Outcomes Measurement Information System (PROMIS®) Cognitive Function- Short Form 4a | In the past 7 days
  The PROMIS® v2.0 Cognitive Function short forms measure participants' subjectively experienced cognitive functioning. Individuals may select one of five options in response: "5-never," "4-rarely (once)," "3-sometimes (2-3 times)," "2-often (about once a day)," and "1-very often (several times a day)." PROMIS scales are expressed on a T score, where 50 is the mean of the general population, with a standard deviation of 10 by definition. Most scores fall between 20 and 80, +/- 3 SDs around the mean. Higher scores represent more of a domain. Lower raw scores and lower T scores on this measure indicate greater subjective cognitive difficulty.
The Patient Feedback Survey | Immediate - This questionnaire is about survey burden in regard to the study
  The Patient Feedback Survey is a brief six-item PRO measure that captures how the patient perceives PROMs administered in terms of burdensomeness. A composite score is calculated to create a weighted representative index of concern, comfort, and well-being relative to time to completion for a range of 0 to 72, with higher scores indicative of elevated endorsed response burden.

CONTACTS AND LOCATIONS:
Overall Officials: James W. Griffith, PhD, Principal Investigator — University of Chicago; Alexander P. Glaser, MD, Principal Investigator — NorthShore University HealthSystem, Department of Surgery, Division of Urology; Abigail R. Smith, PhD, Principal Investigator — Northwestern University
Locations (1):
- NorthShore University HealthSystem Research Institute, Glenview, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data may be shared with other researchers.

REFERENCES:
- [Background] Glaser AP, Smith AR, Maglaque D, Helfand BT, Mohamed R, An H, Marquez M, Talaty P, Carolan P, Geller AM, Farina FR, Jensen SE, Griffith JW. Enhanced clinical decisions for management of benign prostatic hyperplasia using patient-reported outcomes: protocol for a prospective observational study. BMC Urol. 2024 May 21;24(1):110. doi: 10.1186/s12894-024-01500-0. PMID 38773430
- [Derived] Glaser AP, Smith AR, Maglaque D, Helfand BT, Mohamed R, An H, Marquez M, Talaty P, Carolan P, Geller AM, Farina FR, Jensen SE, Griffith JW. Enhanced Clinical Decisions for Management of Benign Prostatic Hyperplasia using Patient-Reported Outcomes: Protocol for a Prospective Observational Study. Res Sq [Preprint]. 2024 May 6:rs.3.rs-4308293. doi: 10.21203/rs.3.rs-4308293/v1. PMID 38766034
- See also: This protocol outlines the rationale and methods to: (1) integrate PROs for better BPH care; (2) assess psychometric properties of the LURN SIs; and (3) develop care-coordination recomm — https://bmcurol.biomedcentral.com/articles/10.1186/s12894-024-01500-0

DOCUMENTS (1):
  • Study Protocol (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/32/NCT05898932/Prot_005.pdf